CLINICAL TRIAL: NCT05454891
Title: Postprandial Glucose Control Using an Extended Bolus for High-fat High Protein Meals in a Closed-loop System in Patients With Type 1 Diabetes
Brief Title: Extended Bolus for Meals in a Closed-loop System
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 58992; 5K23DK121942-02 (NIH)
Record Dates: First submitted 2022-06-24; First posted 2022-07-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned (1:1) in blocks of two to the order in which they receive the two premeal insulin boluses: extended followed by standard bolus or a standard followed by extended bolus.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- High Fat High Protein (HFHP) Meal- extended then standard insulin bolus arm (Experimental): Subjects will receive extended meal bolus for breakfast on the first day and standard meal bolus on the second day of the study.
  Interventions: Drug: Extended bolus of insulin then standard bolus of insulin
- High Fat High Protein (HFHP) Meal- standard then extended insulin bolus arm (Experimental): Subjects will receive standard meal bolus for breakfast on the first day and extended meal bolus on the second day.
  Interventions: Drug: Standard bolus of insulin then extended bolus of insulin

INTERVENTIONS:
Drug: Extended bolus of insulin then standard bolus of insulin — For a standardized HFHP breakfast, participants will receive an extended meal bolus of insulin on the first morning and a standard meal bolus of insulin on the second morning of the study.
  Arms: High Fat High Protein (HFHP) Meal- extended then standard insulin bolus arm
Drug: Standard bolus of insulin then extended bolus of insulin — For a standardized HFHP breakfast, participants will receive a standard bolus of insulin on the first morning and an extended bolus of insulin on the second morning of the study.
  Arms: High Fat High Protein (HFHP) Meal- standard then extended insulin bolus arm

SUMMARY:
This study aims to evaluate whether the use of an extended bolus will improve glucose control with high-fat high protein meals using a closed-loop system. The new knowledge gained from this study may provide a method to allow for the proper administration of insulin over an extended period to mitigate the risk of prolonged hyperglycemia or early hypoglycemia.

ELIGIBILITY:
Inclusion Criteria

* Age between 13 and 19 years old, A1C > 6% at screening
* Diagnosed with type 1 diabetes for at least one year
* Total daily dose (TDD) of insulin ≥ 0.3 units/kg/day
* Currently using the Control IQ closed-loop system
* Willing to abide by meal recommendations and study procedures
* Willing and able to sign the Informed Consent Form (ICF) and/or has a parent or guardian willing and able to sign the ICF
* Use an Android or Apple smartphone
* Willingness not to start any new non-insulin glucose-lowering agent during the course of the trial
* Participant and parent(s)/guardian(s) willingness to participate in all training sessions as directed by study staff
* Parent/guardian proficient in reading and writing English
* Live in the United States, with no plans to move outside the United States during the study period

Exclusion Criteria

* A1C >10%
* One or more episodes of severe hypoglycemia or DKA requiring ER visit or hospitalization within the past three months
* Used non-insulin anti-diabetic medication within the last 30 days other than metformin
* Known history of gastroparesis, seizure disorder, adrenal insufficiency, or ongoing renal or hepatic disease
* Pregnancy or lactation
* Untreated or unstable hypothyroidism
* Currently undergoing cancer treatment or systemic treatment with steroids
* Untreated or inadequately treated mental illness
* Current alcohol abuse
* Current illness that would interfere with participation in the study
* Delayed gastric emptying or any concurrent conditions that can be associated with delayed gastric emptying or altered digestion; and the use of any medication that affects gastric emptying
* Celiac Disease

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Glucose Area Under Curve [AUC] | Baseline and 5 hours post-bolus
  Area under the curve between glucose trace and starting glucose (mg/dL* hour)

SECONDARY OUTCOMES:
Percentage of time between 70-180 mg/dL | Baseline and 5 hours post-bolus
  Percentage of time spent between 70-180 mg/dl based on Continuous Glucose Monitor (CGM) values
Percentage of time in hypoglycemic range (defined as < 70 mg/dL) | Baseline and 5 hours post-bolus
  Percentage of time spent with blood sugar less than 70 mg/dL based on Continuous Glucose Monitor (CGM) values
Average glucose | Baseline and 5 hours post-bolus
  Average glucose value based on Continuous Glucose Monitor (CGM) values
Percentage of time in hyperglycemic range (defined as ≥180 mg/dL); | Baseline and 5 hours post-bolus
  Percentage of time spent with blood sugar higher than 180 mg/dL based on Continuous Glucose Monitor (CGM) values
Insulin dosage | Baseline and 5 hours post-bolus
  Total insulin received during 5 hrs ( manual bolus as well as automated)
Time to target | Baseline and 5 hours post-bolus
  Time spent till blood glucose returns to range
Time to baseline | Baseline and 5 hours post-bolus
  Time spent till blood glucose returns to baseline
Time to peak glucose | Baseline and 5 hours post-bolus
  Time spent till blood glucose reaches the maximum value after meal
Change in glucose | Baseline and 5 hours post-bolus
  The difference between baseline to max glucose value
Peak glucose concentration | Baseline and 5 hours post-bolus
  Max blood glucose
Percentage of time between 70-140 mg/dL | Baseline and 5 hours post-bolus
  Percent of glucose readings from CGM system between 70-140 mg/dL per unit of time

CONTACTS AND LOCATIONS:
Overall Officials: Laya Ekhlaspour, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No